CLINICAL TRIAL: NCT04047511
Title: Immersive Virtual Therapy as a Method Supporting the Non-Farmacological Treatment of Late-Life Depression
Brief Title: Virtual Therapy as a Method Supporting Treatment of Late-Life Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wroclaw University of Health and Sport Sciences (Other)
Collaborators: Foundation for Senior Citizen Activation SIWY DYM (Other)
Responsible Party: Principal Investigator, Błażej Cieślik, Research Assistant, Wroclaw University of Health and Sport Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 59/0203/S/02
Record Dates: First submitted 2019-07-31; First posted 2019-08-06 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Depressive Symptoms; Depression; Anxiety
Keywords: virtual reality; depression; anxiety; mental health; elderly; psychotherapy; rehabilitation
MeSH Terms: conditions — Depression; Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (Experimental): Twice a week, for a 4 consecutive weeks:
  * 8 sessions of VRTierOne therapy ( 20 minutes each)
  * 8 sessions of general fitness training (40 minutes each)
  Interventions: Device: VRTierOne; Behavioral: Group general fitness training
- Control (Active Comparator): Twice a week, for a 4 consecutive weeks:
  * 8 sessions of group psychoeducation and relaxation (20 minutes each)
  * 8 sessions of general fitness training (40 minutes each)
  Interventions: Behavioral: Group general fitness training; Behavioral: Group Psychoeducation

INTERVENTIONS:
Device: VRTierOne — As a virtual reality source, VRTierOne device (Stolgraf®) were used. Thanks to using head mounted display and the phenomenon of total immersion "VRTierOne" Stolgraf® provides an intense visual, auditory and kinesthetic stimulation. It can have a calming and mood-improving effect or help the patients recognize their psychological resources and motivate to the rehabilitation process. In the virtual therapeutic garden there are a rich set of symbols and metaphors based on Ericksonian Psychotherapy approach. The most important is the Garden of Revival which symbolizes the patient's health. It used to be full of life and energy, now it is neglected, requires work to be revived. In the therapeutic process day by day, the lector (therapist) tells the patient a symbolic story about his/her situation. By performing tasks in the virtual garden, the patient influences the course of this story, becomes an active participant of the therapeutic process and sees the effects his work.
  Arms: Virtual Reality
Behavioral: Group general fitness training — A single session of general fitness training will be composed of low-intensity, general-fitness exercises. Most of the exercises will be carried out in a sitting position and standing positon. The session will contain aerobic (general warm-up), musculo-articular (strengthening muscles and joints range of motion) and stabilizing exercises (improve spatio-visual coordination). Perception of effort will be monitored using the Borg 6-20 rating the perceived exertion. Conducted by a physiotherapist in group form.
Behavioral: Group Psychoeducation — A single sesstion will contain mini-lectures about mental well-being and psychohygiene, conduced by a psychotherapist in group form.
  Arms: Control

SUMMARY:
This study evaluates the addition of virtual therapy intervention in the treatment of depression in the elderly. Half of the participants will receive virtual reality treatment as an addition to physical exercises and psychoeducation, while the other half will receive physical exercises and psychoeducation alone.

DETAILED DESCRIPTION:
Depressive disorders are frequent and can either first be manifested at a younger age and recurrent during later life or have an onset beyond 60 years (late-life depression). The multifactorial genesis of depression in old age includes psychosocial, vascular and metabolic factors and requires multimodal and multi-professional therapy including physical activity and psychosocial interventions. However, there is still a percentage of older people who do not show improvement in depressive symptoms.

In recent years, various types of virtual reality are gaining in popularity, primarily because of the availability and ease of use. A systematic review from 2018 concluded that VR treatment had moderate to large effects in anxiety and depression, compared to controls and it could be another effective choice available to clinicians and patients.

Therefore, the aim of this project was to evaluate the effectiveness of virtual therapy in the elderly, in whom the previous multimodal therapeutic program has not brought the expected results.

ELIGIBILITY:
Inclusion Criteria:

* GDS≥10 or HADS-A≥8 or HADS-D≥8

Exclusion Criteria:

* cognitive impairment (MMSE<24) or aphasia and a serious loss of sight or hearing that makes it impossible to assess cognitive functions based on MMSE;
* contraindications for virtual therapy (epilepsy, vertigo, eyesight impairment);
* substance abuse;
* participation in another therapeutic project or individual psychotherapy;
* antidepressant treatment;

Ages: 60 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
The Geriatric Depression Scale (GDS) | 15 minutes
  The Geriatric Depression Scale is a self-report 30-items measure of well-being and mood in older adults. The patient responds in a "Yes/No" format. Scoring ranges from 0 to 30, where 11 and more means mood disorders. The higher score means the greater depression.

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | 30 minutes
  The Hospital Anxiety and Depression Scale (HADS) is a fourteen-item scale scoring from 0 to 3 for each item. The first seven items relate to anxiety (HADS-A), and the remaining seven items relate to depression (HADS-D). The global scoring ranges from 0 to 42 with a cut-off point of 8/21 for anxiety and 8/21 for depression. The higher the score, the greater anxiety or depression symptoms.
Perception of Stress Questionnaire (PSQ) | 30 minutes
  The Perception of Stress Questionnaire (PSQ) is a 27-item scale scoring from 1 to 5 for each item. 21 items examine the level of stress in the area of emotional tension, external stress and intrapsychic stress, and 6 items refer to the lie scale. The global scoring for perception of stress ranges from 21 to 105 with a cut-off point of 60 for high level of perceived stress. The higher the score, the greater the sense of stress. PSQ will be performed at the beginning and after four weeks of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Szczepańska-Gieracha, Professor, Study Director — University School of Physical Education, Wroclaw, Poland; Błażej Cieślik, MSc, Principal Investigator — University School of Physical Education, Wroclaw, Poland
Locations (1):
- Foundation for Senior Citizen Activation SIWY DYM, Wroclaw, Lower Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Valmaggia LR, Latif L, Kempton MJ, Rus-Calafell M. Virtual reality in the psychological treatment for mental health problems: An systematic review of recent evidence. Psychiatry Res. 2016 Feb 28;236:189-195. doi: 10.1016/j.psychres.2016.01.015. Epub 2016 Jan 12. PMID 26795129
- [Background] Freeman D, Reeve S, Robinson A, Ehlers A, Clark D, Spanlang B, Slater M. Virtual reality in the assessment, understanding, and treatment of mental health disorders. Psychol Med. 2017 Oct;47(14):2393-2400. doi: 10.1017/S003329171700040X. Epub 2017 Mar 22. PMID 28325167
- [Background] Maples-Keller JL, Bunnell BE, Kim SJ, Rothbaum BO. The Use of Virtual Reality Technology in the Treatment of Anxiety and Other Psychiatric Disorders. Harv Rev Psychiatry. 2017 May/Jun;25(3):103-113. doi: 10.1097/HRP.0000000000000138. PMID 28475502
- [Background] McCann RA, Armstrong CM, Skopp NA, Edwards-Stewart A, Smolenski DJ, June JD, Metzger-Abamukong M, Reger GM. Virtual reality exposure therapy for the treatment of anxiety disorders: an evaluation of research quality. J Anxiety Disord. 2014 Aug;28(6):625-31. doi: 10.1016/j.janxdis.2014.05.010. Epub 2014 Jun 7. PMID 25093964
- [Background] Li J, Theng YL, Foo S. Game-based digital interventions for depression therapy: a systematic review and meta-analysis. Cyberpsychol Behav Soc Netw. 2014 Aug;17(8):519-27. doi: 10.1089/cyber.2013.0481. Epub 2014 May 8. PMID 24810933